CLINICAL TRIAL: NCT01315899
Title: Phase IIa Study of the Efficacy of ORM-12471 for Prevention of Cold-induced Vasospasm: a Randomised, Double-blind, Placebo-controlled, Single Centre Crossover Study in Patients With Raynaud's Phenomenon Secondary to Systemic Sclerosis
Brief Title: Efficacy of ORM-12741 for Prevention of Raynaud's Phenomenon
Acronym: REINO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommendation by study DSMC to the sponsor following interim analysis of 8 subjects.
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 3098009
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Raynaud's Phenomenon
Keywords: Raynaud's phenomenon; Systemic sclerosis
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ORM-12471 30mg (Experimental)
  Interventions: Drug: ORM-12471 30mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- ORM-12471 100mg (Experimental)
  Interventions: Drug: ORM-12471

INTERVENTIONS:
Drug: ORM-12471 30mg — Given as a single dose once during the crossover study as per Williams design
  Arms: ORM-12471 30mg
Drug: ORM-12471 — Given as a single dose once during the study as per Williams crossover design
  Arms: ORM-12471 100mg
Drug: placebo — Given once as a single dose during the study as per Williams crossover design
  Arms: placebo

SUMMARY:
Raynaud's phenomenon (RP) is a disorder of the digital blood vessels resulting in episodic impairment of blood flow. During an attack of RP which commonly affects the hands and feet these arteries contract briefly which limits the blood flow (this is called a vasospasm) and deprived of blood the skin turns white then blue. The aim of this study is to prove the concept that ORM-12741 can prevent these blood vessel spasms.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Age of 10-75 years (inclusive)
* Body mass index (BMI) between 10-30 kg/m2 (inclusive)
* Male or female patients with a diagnosis of active Raynaud's phenomenon (RP) secondary to systemic sclerosis. Active RP will be defined as a history of cold sensitivity associated with colour changes of cyanosis or pallor, as well as of at least 6 attacks weekly during the winter months. Diagnosis of systemic sclerosis will be defined by the European League Against Rheumatism (EULAR) criteria.
* Stable symptoms for RP and medication requirements within 2 months prior to screening
* Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Treatment with nitrates
* Treatment with calcium channel blockers (CCBs)for indications other than the relief of RP symptoms
* Treatment with calcium channel blockers (CCBs) for the relief of RP symptoms that in the opinion of the investigator cannot be stopped from the screening visit until end of the last experimental session
* Changes in dosing of other vasoactive medications within 1 month prior to screening or during the study
* Smoking or smoking cessation using nicotine products within 3 months prior to screening
* Current active ischemic digital ulcer and/or tissue gangrene
* History of sympathectomy
* Upper extremity deep vein thrombosis or lymphoedema within 3 months prior to screening.
* Clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, neurological, psychiatric or malignant disorder or any other major concurrent illness that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part in the study
* Supine Heart rate (HR) >100 beats per minute (bpm) after a 10 minute rest at screening
* Supine systolic BP (SBP)>160 or diastolic BP (DBP)>100 mmmHg after a 10 minute rest at screening visit
* Any other abnormal value of laboratory, vital signs or ECG which may in the opinion of the investigator interfere with the interpretation of the study results or cause a health risk for the subject if he/she takes part into the study.
* Pregnant or breast feeding or considering pregnancy in the next 4 months
* Female subjects of child bearing potential (i.e. menstruating or less than 2 years post menopausal) if they are not using proper contraception (hormonal contraception,intrauterine device [IUD] or surgical sterilisation, spermicidal foam in conjunction with condom on male partner)
* Subjects with pre-planned elective surgery during the estimated study period
* Blood donation or loss of a significant amount of blood within 30 days prior to screening
* Participation in a drug study within 30 days prior to screening
* Known hypersensitivity to the active substance or to any excipients of the drug
* Recent or current (suspected) drug abuse
* Recent or current alcohol abuse (regular drinking more than 14 units per week for females or 21 units per week for males 1 unit= 4cl of spirits or equivalent)
* Inability to refrain from consuming caffeine-containing beverages for at least 12 hours prior to and during treatment visits e.g propensity in getting headache when refraining from caffeine-containing beverages
* Inability to participate in all treatment periods
* Unsuitable veins for repeated venipuncture or for cannulation
* The subject is not able to swallow a test capsule at the screening visit
* Any other condition that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the patient if he/she takes part in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Finger temperature measurements and laser doppler imaging of the hands | 0-90minutes continuous measurement
  Finger temperature measurements and laser doppler imaging of the hands will be continually monitored from 0 minutes through to 90 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane L Herrick, MB,ChB, MD, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Salford Royal NHS foundation Trust, Salford, Greater Manchester, United Kingdom

REFERENCES:
- [Result] Herrick AL, Murray AK, Ruck A, Rouru J, Moore TL, Whiteside J, Hakulinen P, Wigley F, Snapir A. A double-blind, randomized, placebo-controlled crossover trial of the alpha2C-adrenoceptor antagonist ORM-12741 for prevention of cold-induced vasospasm in patients with systemic sclerosis. Rheumatology (Oxford). 2014 May;53(5):948-52. doi: 10.1093/rheumatology/ket421. Epub 2014 Jan 31. PMID 24489014